CLINICAL TRIAL: NCT05881720
Title: Effect of Sacubitril/Valsartan Versus Valsartan on Left Ventricular Ejection Fraction and Biomarker in Heart Failure
Brief Title: Sacubitril/Valsartan Versus Valsartan in Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sacubitril/valsartan in HF
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure
Keywords: LVEF%,; Lipo A,; troponin I,; NT-Pro BNP,; neopterin
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; sacubitril; Valsartan

STUDY DESIGN:
Intervention Model Description: Group 1 (N = 40) received sacubitril/valsartan (target dose, 100 mg twice daily) or group 2 received valsartan (target dose, 80 mg twice daily) in addition to recommended therapy according to physician's judgment.
Who Masked: Participant, Investigator
Masking Description: Double Blind randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (N = 40) (Experimental): Group 1 (N = 40) received sacubitril/valsartan (target dose, 100 mg twice daily) in addition to recommended therapy according to physician's judgment.
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet
- Group 2 (N = 40) (Experimental): group 2 received valsartan (target dose, 80 mg twice daily) in addition to recommended therapy according to physician's judgment.
  Interventions: Drug: Valsartan 80 mg

INTERVENTIONS:
Drug: Sacubitril / Valsartan Oral Tablet — Group 1 (N = 40) received sacubitril/valsartan (target dose, 100 mg twice daily) in addition to recommended therapy according to physician's judgment.
  Other Names: sacubitril / valsartan (100 mg twice daily)
  Arms: Group 1 (N = 40)
Drug: Valsartan 80 mg — group 2 received valsartan (N=40, target dose, 80 mg twice daily) in addition to recommended therapy according to physician's judgment.
  Other Names: Valsartan
  Arms: Group 2 (N = 40)

SUMMARY:
The objective of this study was to identify potential prognostic factors of sacubitril/valsartan vs Valsartan treatment response.

DETAILED DESCRIPTION:
Study will include 80 symptomatic patients with chronic HFrEF (left ventricular ejection fraction ≤35%) and New York Heart Association (NYHA) class II/III: Group 1 (N = 40) received sacubitril/valsartan (target dose, 100 mg twice daily) or group 2 received valsartan (target dose, 80 mg twice daily) in addition to recommended therapy according to physician's judgment. Analysis of biochemical parameters, cardiopulmonary exercise testing, and echocardiographic evaluation was performed at baseline and 6 months later. The primary outcome was the change in LVEF%, Lipo A, troponin I, NT-Pro BNP and neopterin levels. The secondary outcome is reporting efficacy and safety of sacubitril/valsartan vs Valsartan use and the relationship between NYHA and EF and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HF were enrolled if aged > 35 years,
* Stable symptomatic systolic chronic HF (≥ 4 weeks), with left ventricular ejection fraction (LVEF) < 35%,
* NYHA class II-III,
* Sinus rhythm and resting HR ≥ 70 beats/min on optimised standard medical therapy.

Exclusion Criteria:

* Patients with acute decompensation,
* Cerebrovascular events during the previous 6 months,
* Pregnancy, breastfeeding,
* Any valve dysfunction/abnormality,
* Active myocarditis,
* Second-degree and third-degree atrioventricular block,
* Sick sinus syndrome.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
LVEF % | 6 months
  left ventricular ejection fraction percent
Lipo A (pg/ml) | 6 months
  Lipo protien A (pg/ml)
Troponin.I (ng/ml) | 6 months
  Troponin.I (ng/ml) biomarker
NT-Pro BNP | 6 months
  NT-pro BNP(pg/ml) biomarker
Neopterin (nmol/l) | 6 Months
  Neopterin biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass.Prof., Study Chair — Damanhour University; Ahmed El-Sherbeni, Study Director — Tanta University; Lamiaa Khedr, Principal Investigator — Tanta University
Locations (1):
- Tanta University Hospital, Tanta, Elgarbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dogheim GM, Khairat I, Omran GA, El-Haggar SM, Amrawy AME, Werida RH. Clinical comparative study assessing the effect of ivabradine on neopterin and NT-Pro BNP against standard treatment in chronic heart failure patients. Eur J Clin Pharmacol. 2022 Jun;78(6):943-954. doi: 10.1007/s00228-022-03290-6. Epub 2022 Mar 3. PMID 35238960
- [Background] McMurray JJV, Jackson AM, Lam CSP, Redfield MM, Anand IS, Ge J, Lefkowitz MP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Rizkala AR, Sabarwal SV, Shah AM, Shah SJ, Shi VC, van Veldhuisen DJ, Zannad F, Zile MR, Cikes M, Goncalvesova E, Katova T, Kosztin A, Lelonek M, Sweitzer N, Vardeny O, Claggett B, Jhund PS, Solomon SD. Effects of Sacubitril-Valsartan Versus Valsartan in Women Compared With Men With Heart Failure and Preserved Ejection Fraction: Insights From PARAGON-HF. Circulation. 2020 Feb 4;141(5):338-351. doi: 10.1161/CIRCULATIONAHA.119.044491. Epub 2019 Nov 17. PMID 31736337
- [Background] Biering-Sorensen T, Lassen MCH, Shah A, Claggett B, Zile M, Pieske B, Pieske-Kraigher E, Voors A, Shi V, Lefkowitz M, Packer M, McMurray JJV, Solomon SD; PARAMOUNT Investigators. The Effect of Sacubitril/Valsartan on Left Ventricular Myocardial Deformation in Heart Failure with Preserved Ejection Fraction (PARAMOUNT trial). J Card Fail. 2023 Jun;29(6):968-973. doi: 10.1016/j.cardfail.2023.03.019. Epub 2023 Apr 7. PMID 37031887